CLINICAL TRIAL: NCT04555525
Title: A Pilot Study on the Use of Seysara for Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Responsible Party: Principal Investigator, L.H. Kircik, M.D., Medical Director, Derm Research, PLLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEY1901
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Results first posted 2020-12-16 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Acne Rosacea
MeSH Terms: conditions — Rosacea | interventions — sarecycline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sarecycline (Experimental): weight-based dose per label by mouth once daily for 12 weeks
  Interventions: Drug: sarecycline
- Centrum Adult Multivitamin (Other): one tablet by mouth daily for 12 weeks
  Interventions: Dietary Supplement: Centrum Adult Multivitamin

INTERVENTIONS:
Drug: sarecycline — sarecycline tablet
  Other Names: Seysara; sarecycline hydrochloride
  Arms: sarecycline
Dietary Supplement: Centrum Adult Multivitamin — Centrum Adult Mulltivitamin tablet
  Arms: Centrum Adult Multivitamin

SUMMARY:
This is a prospective, parallel group, randomized, investigator-blinded pilot study. Approximately 100 subjects will be randomized at a 3:1 ratio to Seysara (sarecycline) at a weight-based dose per label or Centrum Adult Multivitamin to take by mouth daily. The study is comprised of 5 visits: screening, baseline, week 4, week 8, and week 12. Investigators will perform rosacea IGA (Investigator Global Assessment,) inflammatory lesion count, record adverse events and con meds, and ask each subject to complete a DLQI (Dermatology Life Quality Index.)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Moderate to severe rosacea (IGA score 3 or 4) on the proposed facial treatment area consisting of:

   1. At least 15 and not more than 50 facial papules and pustules, excluding lesions involving the eyes and scalp
   2. No more than 2 nodules on the face
3. Presence or history of erythema and/or flushing of the face
4. If a female of child-bearing potential, have a negative urine pregnancy test and agree to use an effective method of contraception. A sterile sexual partner is NOT considered an adequate form of birth control
5. Willing to minimize external factors that might trigger rosacea flare-ups (eg, spicy foods, thermally hot foods and drinks, hot environments, prolonged sun exposure, strong winds, and alcoholic beverages
6. Subjects who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to use the same make-up, brand/type, or frequency of use throughout the study
7. Completed and signed an appropriately administered Informed Consent Form (ICF) prior to any study-related procedures -

Exclusion Criteria:

1. Woman who is pregnant, lactating, or planning to become pregnant during the study period
2. presence of any skin condition on the face that would interfere with the diagnosis or assessment of rosacea
3. Moderate or severe rhinophyma, dense telangiectasia (score 3, severe;) or plaque-like facial edema
4. Excessive facial hair (eg, beards, sideburns, moustaches, etc) that would interfere with diagnosis or assessment of rosacea
5. History of hypersensitivity or allergy to all tetracyclines, or to any other component of the formulation
6. Patients with history of C-diff associated colitis, intracranial hypertension will be excluded
7. Severe erythema, dryness, scaling, pruritis, stinging/burning, or edema
8. Use within 6 months prior to Day 0/Baseline of oral retinoids (eg, Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed)
9. Initiation of use of estrogens or oral contraceptives less than 3 months prior to Day 0/Baseline
10. Use within 1 month prior to Day 0/Baseline of:

    1. Systemic antibiotics known to have an impact on the severity of facial rosacea (eg, containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim.) Subjects requiring systemic antibiotics not known to affect rosacea will be considered on a case-by-case basis
    2. Systemic corticosteroids (Note: intranasal and inhalational corticosteroids do not require a washout and maybe used throughout the trial if the subject is on a stable dose.)
11. Use within 2 weeks prior to Day 0/Baseline of:

    1. Topical corticosteroids
    2. Topical antibiotics
    3. Topical medications for rosacea (eg, metronidazole)
12. Use of sauna during the 2 weeks prior to Day 0/Baseline and during the study
13. Had wax epilation of the face within 2 weeks prior to Day 0/Baseline
14. Active bacterial folliculitis
15. Consumption of excessive alcohol, abuse of licit or illicit drugs, or a condition that, in the opinion of the Investigator, could compromise the subject's ability to comply with study requirements
16. Participation in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold
17. Presence of any clinically significant condition or situation, other than the condition being studied, that in the opinion of the Investigator would interfere with the study evaluations or optimal participation in the study
18. Participation in an investigational drug study (ie, subject has been treated with an investigational drug) within 30 days prior to Day 0/Baseline. Subjects who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion
19. Prior laser therapy (for telangiectasia or other conditions), electrodessication, or phototherapy (eg, ClearLight ®) to the facial area within 180 days prior to Day 0/Baseline
20. Prior cosmetic procedures (eg, facials) that may affect the efficacy and safety profile of the investigational product within 14 days prior to Day 0/Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Sciences, PLLC, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Started | 75 | 25
Completed | 72 | 25
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sarecycline | Centrum Adult Multivitamin | Total
Number analyzed (Participants) | 72 | 25 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.42 (14.96) | 52.36 (13.47) | 52.41 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 22 | 80
  Male | 14 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 69 | 25 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 72 | 25 | 97

OUTCOME MEASURES:

1. Primary Outcome: IGA (Investigator Global Assessment)
Description: Percent of subjects achieving clear or almost clear on IGA. The Investigator will score rosacea at each visit as per the following IGA:
  0 = Clear (No inflammatory lesions present, no erythema); 1 = Almost Clear (Very few small papules/pustules, very mild erythema present); 2 Mild (Few small or large papules/pustules, moderate erythema); 3= Moderate (Several small or large papules/pustules, moderate erythema); 4 = Severe (Numerous small and/or large papules/pustules, severe erythema)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Number analyzed (Participants) | 72 | 25
Participants | 54 | 4

2. Primary Outcome: Inflammatory Lesion Count
Description: Change in inflammatory lesion count
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Number analyzed (Participants) | 72 | 25
Percent Change | -80 (24) | -60 (32)

3. Secondary Outcome: IGA
Description: as for outcome 1
Time Frame: week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Number analyzed (Participants) | 72 | 25
Participants | 15 | 2

4. Secondary Outcome: IGA
Description: as for outcome 1
Time Frame: week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Number analyzed (Participants) | 72 | 25
Participants | 32 | 3

5. Secondary Outcome: Inflammatory Lesion Count
Description: Change in inflammatory lesion count
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Number analyzed (Participants) | 72 | 25
Percent Change | -56 (29) | -31 (30)

6. Secondary Outcome: Inflammatory Lesion Count
Description: Change in inflammatory lesion count
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Sarecycline | Centrum Adult Multivitamin
Number analyzed (Participants) | 72 | 25
Percent Change | -71 (27) | -44 (42)

ADVERSE EVENTS:
Time Frame: 12 weeks average, from signing of Informed Consent until end of study participation.
Arm/Group | Sarecycline | Centrum Adult Multivitamin
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/25
Other Adverse Events (participants affected / at risk) | 16/72 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarecycline (N=72) | Centrum Adult Multivitamin (N=25)
Boil (Skin and subcutaneous tissue disorders) | 1 (1) | 0
bone spur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
cholecystectomy (Surgical and medical procedures) | 1 (1) | 0
cholelithiasis worsening (Hepatobiliary disorders) | 1 (1) | 0
dry lips (Skin and subcutaneous tissue disorders) | 1 (1) | 0
facial sunburn (Skin and subcutaneous tissue disorders) | 1 (1) | 0
dog bite r arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0
generalized muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
headache (Nervous system disorders) | 2 (2) | 0
herpes simplex l lower lip (Infections and infestations) | 1 (1) | 0
influenza (Infections and infestations) | 1 (1) | 0
ingrown eyebrow hair (Skin and subcutaneous tissue disorders) | 1 (1) | 0
intermittent pain under r rib cage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
metallic taste (Gastrointestinal disorders) | 1 (1) | 0
nausea (Gastrointestinal disorders) | 1 (1) | 0
r ear infection (Ear and labyrinth disorders) | 1 (1) | 0
rash of unknown origin (Skin and subcutaneous tissue disorders) | 1 (1) | 0
respiratory syncytial virus (Infections and infestations) | 1 (1) | 0
sinus infection (Infections and infestations) | 1 (1) | 0
sleep apnea (Nervous system disorders) | 1 (1) | 0
stomach bloating (Gastrointestinal disorders) | 1 (1) | 0
sunburn on face (Skin and subcutaneous tissue disorders) | 1 (1) | 0
tinea versicolor (Infections and infestations) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT04555525/Prot_SAP_000.pdf